CLINICAL TRIAL: NCT06110364
Title: Vagal Nerve Stimulation as an Alternative Therapy for Premature Ventricular Contractions
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study Closed due to funding; no subjects enrolled
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Principal Investigator, Jose Huizar, Associate Chief of Staff for Research and Development at VAMC, Professor of Medicine at VCU, Director, Arrhythmia and Device Clinic at VAMC and Affiliate Professor of Physiology and Biophysics VCU, Hunter Holmes Mcguire Veteran Affairs Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1724039
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Premature Ventricular Contraction
Keywords: NIVNS Non-invasive vagal nerve stimulation; LLTS- Low-level tragus stimulation; HRV-BF - Heart rate variability biofeedback
MeSH Terms: conditions — Ventricular Premature Complexes | interventions — Transcutaneous Electric Nerve Stimulation; Breathing Exercises

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to Premature ventricular contraction suppression strategies: 1) Lower level tragus stimulation 2) Heart rate variability biofeedback and 3) conventional medical therapy (usual care)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Low-Level Tragus Stimulation (Experimental): The Low-Level Tragus Stimulation will be done with TENS.
  Interventions: Device: Low-Level Tragus Stimulation
- Heart Rate Variability- Biofeedback (Experimental): Heart Rate Variability-Biofeedback will be done with a phone application. Practice sessions are at least 10-15 minutes twice a daily.
  Interventions: Behavioral: Heart Rate Variability- Biofeedback
- Conventional Medical Therapy (Active Comparator): Subjects without beta blockers will be initiated on a usual/standard care medication of beta blockers to determine the efficacy of this standard medication therapy for Premature Ventricular Contraction suppression.
  Interventions: Other: Conventional Medical Therapy

INTERVENTIONS:
Device: Low-Level Tragus Stimulation — Low-Level Tragus Stimulation via TENS unit will be monitored with a Holter.
  Other Names: TENS
  Arms: Low-Level Tragus Stimulation
Behavioral: Heart Rate Variability- Biofeedback — Heart Rate Variability- Biofeedback will be monitored with a Holter.
  Other Names: Breathing Exercises / Inner Balance
  Arms: Heart Rate Variability- Biofeedback
Other: Conventional Medical Therapy — Conventional Medical Therapy by Beta Blockers will be added to subjects usual care by their doctor if they are not already taking this medication.
  Other Names: Usual care medication
  Arms: Conventional Medical Therapy

SUMMARY:
Prospective randomized control pilot study

DETAILED DESCRIPTION:
The primary aims of this investigator initiated study is :

Aim 1: to assess the ability of non-invasive vagal nerve stimulation to suppress Premature Ventricular Contractions and Aim 2: to compare the efficacy of Lower-level Tragus stimulation and Heart rate variability- Biofeedback in suppression of Premature Ventricular Contractions.

ELIGIBILITY:
Inclusion Criteria:

* Normal Left Ventricular systolic function
* Frequent PVCs

Exclusion Criteria:

* Current use of any (I and/or III) antiarrhythmic medication
* Contraindication to use beta blockers and non-dihydropyridine calcium channel blockers
* Complete Atrioventricular block and pacemaker dependent
* Ongoing uncontrolled hypertension with systolic Blood Pressure> 180
* Family history of dilated Cardiomyopathy in a first degree relative
* Alcohol use disorder or illicit drug use
* Actively being treated Atrial fibrillation/ Flutter with Rapid Ventricular Response
* Moderate to severe valve disorders
* Patient with shortwave/microwave therapy equipment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Assess the ability of non-invasive vagal nerve stimulation to suppress Premature Ventricular Contractions. | perspective 12-week study (each arm lasting two weeks with a one week washout between each arm)
  Compare the effects of Premature Ventricular Contractions suppression between standard medical therapy and non-invasive vagal nerve stimulation.

SECONDARY OUTCOMES:
Compare the efficacy of non-invasive vagal nerve stimulation via lower-level vagal stimulation and heart rate variability in suppression of Premature Ventricular Contractions. | perspective 12-week study (each arm lasting two weeks with a one-week washout between each arm)
  It is speculated that Heart Rate Variability-Biofeedback is as effective as Lower Level Tragus Stimulation to achieve successful Premature Ventricular Contraction suppression.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Huizar, M.D., Principal Investigator — Hunter Holmes McGuire Veterans Medical Center
Locations (1):
- Richmond VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Premature ventricular contractions activate vagal afferents and alter autonomic tone: implications for premature ventricular contraction-induced cardiomyopathy — https://pubmed.ncbi.nlm.nih.gov/31322427/
- See also: Relationship between burden of premature ventricular complexes and left ventricular function — https://pubmed.ncbi.nlm.nih.gov/20348027/
- See also: Clinical and translational insights on premature ventricular contractions and PVC-induced cardiomyopathy — https://pubmed.ncbi.nlm.nih.gov/33857575/
- See also: Evaluation and management of premature ventricular complexes — https://pubmed.ncbi.nlm.nih.gov/23733905/
- See also: Stellate ganglion blockade and bilateral cardiac sympathetic denervation in patients with life-threatening ventricular arrhythmias — http://pubmed.ncbi.nlm.nih.gov/28471068/
- See also: Cardiac Sympathetic Denervation for Refractory Ventricular Arrhythmias — https://pubmed.ncbi.nlm.nih.gov/28641796/
- See also: TREAT AF (Transcutaneous Electrical Vagus Nerve Stimulation to Suppress Atrial Fibrillation): A Randomized Clinical Trial — https://pubmed.ncbi.nlm.nih.gov/32192678/
- See also: Heart rate variability biofeedback based on slow-paced breathing with immersive virtual reality nature scenery. — http://pubmed.ncbi.nlm.nih.gov/31616353/
- See also: Non-invasive low-level tragus stimulation in cardiovascular diseases — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC7330730/
- See also: Critical Review of Transcutaneous Vagus Nerve Stimulation: Challenges for Translation to Clinical Practice — http://pubmed.ncbi.nlm.nih.gov/32410932/

DOCUMENTS (1):
  • Informed Consent Form (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT06110364/ICF_000.pdf